CLINICAL TRIAL: NCT02603328
Title: Phase I-II Randomized, Placebo-Controlled, Single-Blinded, Single-Site Clinical Trial of Atorvastatin in the Treatment of Cavernous Angiomas With Symptomatic Hemorrhage Exploratory Proof of Concept (AT CASH EPOC)
Brief Title: Atorvastatin Treatment of Cavernous Angiomas With Symptomatic Hemorrhage Exploratory Proof of Concept (AT CASH EPOC) Trial
Acronym: AT CASH EPOC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB18-0445
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Cavernous Malformation
Keywords: Cerebral cavernous malformation; Statins; MRI; Permeability; Quantitative susceptibility mapping
MeSH Terms: conditions — Hemangioma, Cavernous, Central Nervous System | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator): Atorvastatin 80mg OD (optimal dose). Treatment dose will be de-escalated to 40mg based on reported adverse events.
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): Identically looking capsules containing no active ingredient
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Atorvastatin — 40-80 mg OD
  Arms: Treatment
Other: Placebo — inactive
  Arms: Placebo

SUMMARY:
This phase I/II randomized, placebo-controlled, double-blinded, single-site clinical trial is designed to investigate the effect of a prolonged course of atorvastatin versus placebo on CCM lesional iron deposition assessed by validated quantitative susceptibility mapping (QSM) MRI studies in patients who suffered a symptomatic bleed within the preceding one year.

DETAILED DESCRIPTION:
This phase I/II randomized, placebo-controlled, double-blinded, single-site clinical trial is designed to investigate the effect of a prolonged course of atorvastatin versus placebo on CCM lesional iron deposition assessed by validated quantitative susceptibility mapping (QSM) MRI studies in patients who suffered a symptomatic bleed within the preceding one year. Subjects will also be assessed by lesional and brain vascular permeability MRI using dynamic contrast enhanced quantitative perfusion (DCEQP) and a number of clinical evaluation tools. Subjects shall be followed for 2 years from randomization, the period of highest likelihood of rebleed after a recent CCM hemorrhage. Subjects will undergo clinical and MRI evaluations at baseline, and at 12 and 24 months during the study period. Enrolled subjects and the treating team will be blinded to treatment group allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CCM of any genotype supported by relevant imaging studies.
2. Symptomatic CCM bleeding event within 1 year prior to enrollment.
3. Must be willing/able to travel to the study site for all study visits (baseline, 12 months, and 24 months) over the course of the study period.

Exclusion Criteria:

1. Pre-menopausal women who are breastfeeding, pregnant or likely to get pregnant during the study period.
2. Previous cranial irradiation or surgical/radiosurgical treatment of CCM lesion.
3. Failure to pass MRI safety screening (claustrophobia, metal implant . . . etc)
4. Known allergy or intolerance to gadolinium.
5. Severely impaired renal function (eGFR < 60ml/min), active renal disease or status post-kidney transplants.
6. Statin therapy, for any indication, for more than 7 continuous days or greater than 14 total days within 12 months preceding enrollment.
7. Indication to use statin medication for current approved indication, unrelated to CCM
8. Known allergy or intolerance to statins
9. Liver dysfunction or active liver disease (including chronic viral hepatitis) defined as baseline serum transaminases levels twice the upper range of normal.
10. Previous diagnosis of skeletal muscle disorders of any cause (myopathy), or baseline creatine kinase level five times the upper range of normal.
11. Currently treated with or likely to need treatment with one or more of prohibited medications listed in the protocol.
12. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
13. Serious illness (requiring systemic treatment and/or hospitalization) until subject either completes therapy or is clinically stable on therapy, in the opinion of the site investigator, for at least 30 days prior to study entry.
14. Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated, including conditions resulting in or precipitating myopathy (e.g. HIV, uncontrolled hypothyroidism).
15. In the investigator's opinion, the patient is unstable, and would benefit from a specific intervention rather than treatment with atorvastatin.
16. Inability or unwillingness of subject or legal guardian/representative to give written informed consent.
17. No documentation of valid healthcare insurance.
18. No medical record confirmation of primary care physician.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issam A Awad, MD, Study Chair — Director of Neurovascular Surgery University of Chicago Medicine and Biological Sciences; Daniel F Hanley, MD, Study Chair — Director, Division of Brain Injury Outcomes Service The Johns Hopkins Medical Institutions
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Ali B, Shenkar R, Lee J, Alcazar-Felix RJ, Thompson RE, Stadnik A, Sader G, Polster SP, Flemming KD, Liao JK, Sorrentino M, Girard R, Hanley DF, Awad IA. Recurrent Symptomatic Hemorrhage in Cerebral Cavernous Malformations After Discontinuation of Atorvastatin or Placebo. J Am Heart Assoc. 2026 Jan 29:e46943. doi: 10.1161/JAHA.125.046943. Online ahead of print. PMID 41608890
- [Derived] Alcazar-Felix RJ, Thompson RE, Stadnik A, Kinkade S, Sader G, Jhaveri A, Lee J, Iqbal J, Polster SP, Shenkar R, Flemming KD, Girard R, Carroll TJ, Hanley DF, Awad IA. Relevance of Lesion Volume as an Outcome in Cerebral Cavernous Malformation Drug Trial: Exploratory Analyses in Atorvastatin Treatment of Cavernous Angiomas with Symptomatic Hemorrhage Exploratory Proof of Concept. Neurosurgery. 2025 Oct 21. doi: 10.1227/neu.0000000000003814. Online ahead of print. PMID 41117517
- [Derived] Awad IA, Alcazar-Felix RJ, Stadnik A, Kinkade S, Jhaveri A, Lee J, Hage S, Iqbal J, Polster SP, Shenkar R, Treine K, McBee N, Ostapkovich N, Lane K, Liao JK, Sorrentino M, Lee C, Flemming KD, Girard R, Carroll TJ, Thompson RE, Hanley DF. Safety and efficacy of atorvastatin for rebleeding in cerebral cavernous malformations (AT CASH EPOC): a phase 1/2a, randomised placebo-controlled trial. Lancet Neurol. 2025 Apr;24(4):295-304. doi: 10.1016/S1474-4422(25)00036-5. PMID 40120614

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 80 participants were randomized and followed for 2 years and all results are provided only for these participants.
Groups:
- Treatment 80mg: Atorvastatin 80mg OD (optimal dose). Treatment dose will be de-escalated to 40mg based on reported adverse events.
  Atorvastatin: 40-80 mg OD
Period: Overall Study
Arm/Group | Treatment 80mg | Placebo
Started | 41 | 39
Completed Year 1 | 34 | 36
Lowered to 40mg Dose in Year 1 | 1 | 0
Completed Year 2 | 31 | 31
Lowered to 40mg Dose in Year 2 | 0 | 0
Completed | 31 | 31
Not Completed | 10 | 8

BASELINE CHARACTERISTICS:
Population: Baseline characteristics of intention to treat cohort
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 39 [34 to 54] | 41 [34 to 49] | 41 [34 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 15 | 14 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 34 | 31 | 65
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 32 | 31 | 63
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 2 | 2
Familial cavernous malformation syndrome [Count of Participants; unit: Participants] | 18 | 11 | 29
MRI characteristics - number of lesions [Median (Inter-Quartile Range); unit: Lesions]
  Number of lesions on susceptibility weighted imaging in familial cases | 1 [1 to 13] | 1 [1 to 6] | 1 [1 to 9]
  Number of lesions on T2 ≥4mm in familial cases | 1 [1 to 5] | 1 [1 to 1] | 1 [1 to 3]
Location of index CCM lesion with symptomatic hemorrhage [Number; unit: participants]
  Brainstem | 23 | 21 | 44
  Cerebellum | 2 | 2 | 4
  Frontal Lobe | 3 | 2 | 5
  Occipital Lobe | 1 | 3 | 4
  Parietal Lobe | 1 | 2 | 3
  Temporal Lobe | 2 | 6 | 8
  Thalamus | 5 | 2 | 7
  Other location | 4 | 1 | 5
Time from most recent symptomatic hemorrhage to enrollment, days [Median (Inter-Quartile Range); unit: Days] | 103 [51 to 171] | 104 [69 to 137] | 104 [57 to 150]
Number of symptomatic hemorrhages before enrollment [Median (Inter-Quartile Range); unit: Number of symptomatic hemorrhages] | 1 [1 to 2.50] | 1 [1 to 2] | 1 [1 to 2]
Modified Rankin Scale score [Number; unit: participants] — The mRS (modified Rankin Score) is a simple global measure of functional disability. Scores range from 0 (no symptoms) to 6 (death). An mRS score of 0 to 1 is considered a minimal clinical disability, and 0 to 2 is independent.
  participants
    0 | 6 | 8 | 14
    1 | 18 | 25 | 43
    2-3 | 17 | 6 | 23
    4 | 0 | 0 | 0
    5-6 | 0 | 0 | 0
European quality of life index Visual Analog Scale [Mean (Standard Deviation); unit: units on a scale] — The EQ-VAS (European Quality of Life Visual Analogue Scale) is a vertical visual analogue scale that takes values between 100 (best imaginable health) and 0 (worst imaginable health), on which patients provide a global assessment of their health (patients select how they perceive their current health on a 0 to 100 scale).
  units on a scale | 74.59 (16.29) | 78.28 (12.67) | 76.4 (14.7)
MRI characteristics - size of lesion on T2, mm [Median (Inter-Quartile Range); unit: Size on T2, mm] | 14.70 [9.65 to 18] | 16 [10 to 23.70] | 14.80 [9.75 to 19.80]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Mean Lesional QSM (QSM Change Score)
Description: QSM change score is the Percentage Change in mean lesional iron deposition per year (QSM score) according to assigned treatment (modified intention-to-treat cohort), presented as a mean value across all participants from baseline to year 1 and year 1 to year 2 follow-up MRIs.
  Quantitative susceptibility mapping (QSM) is a noninvasive MRI technique that assesses iron content by quantifying the magnetic susceptibility of local tissues.
  A higher QSM value corresponds to a larger amount of iron in the lesion, which means more blood is present in the lesion.
Time Frame: 2 years of follow-up
Measure: Mean (Standard Error); unit: absolute value of percent change
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 33 | 31
absolute value of percent change
  QSM change score by assigned treatment; year 1 minus baseline | 7.35 (9.77) | 0.24 (10.08)
  QSM change score by assigned treatment; year 2 minus year 1 | 15.18 (10.80) | 26.80 (11.22)

2. Secondary Outcome: Percent Change in Dynamic Contrast-enhanced Quantitative Perfusion (DCEQP) Value (Vascular Permeability) in Index Lesion (Lesional DCEQP Change Score)
Description: DCEQP change score is the absolute value of the Percent Change in DCEQP value of the index lesion, presented as a mean value across all participants from baseline to year 1 and year 1 to year 2 follow-up MRIs
  DCEQP measures vascular permeability and perfusion, in this case as measured in the index lesion. A higher DCEQP value reflects higher permeability in the lesion.
Time Frame: 2 years of follow-up
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 33 | 31
percent change
  Mean lesional DCEQP percent change by assigned treatment; year one minus baseline | 103.40 (40.64) | 35.69 (50.59)
  Mean lesional DCEQP percent change by assigned treatment; year two minus year one | 124.52 (85.15) | 124.82 (88.92)

3. Secondary Outcome: Compare the Changes in Modified Rankin Score Between Atorvastatin and Placebo Groups at the Year 1 Follow-up Visit
Description: Compare the changes in modified Rankin Score between atorvastatin and placebo groups at the year 1 follow-up visit.
  The mRS is a simple global measure of functional disability. Scores range from 0 (no symptoms) to 6 (death). An mRS score of 0 to 1 is considered a minimal clinical disability, and 0 to 2 is independent.
Time Frame: 1 year of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 36
Participants
  mRS 0 | 2 | 8
  mRS 1 | 25 | 20
  mRS 2-3 | 8 | 8
  mRS 4 | 0 | 0
  mRS 5-6 | 0 | 0

4. Secondary Outcome: Compare the Changes in Modified Rankin Score Between Atorvastatin and Placebo Groups at the Year 2 Follow-up Visit.
Description: Compare the changes in modified Rankin Score between atorvastatin and placebo groups at the year 2 follow-up visit (change between mRS score at year 1 follow up visit and year 2 follow up visit).
  The mRS is a simple global measure of functional disability. Scores range from 0 (no symptoms) to 6 (death). An mRS score of 0 to 1 is considered a minimal clinical disability, and 0 to 2 is independent.
Time Frame: 1 year of follow-up (from year 1 to year 2)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 31 | 31
Participants
  mRS 0 | 6 | 12
  mRS 1 | 17 | 12
  mRS 2-3 | 7 | 7
  mRS 4 | 1 | 0
  mRS 5-6 | 0 | 0

5. Secondary Outcome: Mean Score of European Quality of Life Visual Analogue Scale (EQ-VAS) at the Year 1 Follow-up Visit.
Description: Mean score of European Quality of Life Visual Analogue Scale (EQ-VAS) at the year 1 follow-up visit
  The EQ-VAS is a vertical visual analogue scale that takes values between 100 (best imaginable health) and 0 (worst imaginable health), on which patients provide a global assessment of their health.
Time Frame: 1 year of follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 36
score on a scale | 78.3 (17.5) | 78.1 (17.1)

6. Secondary Outcome: Mean Score of European Quality of Life Visual Analogue Scale (EQ-VAS) at the Year 2 Follow-up Visit
Description: Mean score of European Quality of Life Visual Analogue Scale (EQ-VAS) at the year 2 follow-up visit
  The EQ-VAS is a vertical visual analogue scale that takes values between 100 (best imaginable health) and 0 (worst imaginable health), on which patients provide a global assessment of their health.
Time Frame: 1 year of follow up (from year 1 to year 2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 31 | 31
score on a scale | 80.1 (16.0) | 80.5 (12.0)

7. Secondary Outcome: Compare Rate of Drug Compliance in Atorvastatin vs Placebo Group
Description: Compare number of subjects with 90% or greater protocol compliance throughout the 2 year follow-up period
Time Frame: 2 years of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 33 | 31
Participants | 33 | 31

8. Secondary Outcome: Mean Percent Change in Rho-associated Protein Kinase (ROCK) Activity in Peripheral Blood Leukocytes From Baseline to Year 1
Description: Compare the mean percent change in peripheral blood leukocyte ROCK activity between atorvastatin and placebo groups from baseline to year 1
Time Frame: 1 year of follow-up
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 33 | 31
percent change | 32.68 (75.72) | 22.73 (80.21)

9. Secondary Outcome: Mean Percent Change in Rho-associated Protein Kinase (ROCK) Activity in Peripheral Blood Leukocytes From Baseline to Year 2
Description: Compare the mean percent change in peripheral blood leukocyte ROCK activity between atorvastatin and placebo groups from baseline to year 2
Time Frame: 2 year follow-up
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 33 | 31
percent change | 68.17 (101.2) | 55.62 (95.22)

ADVERSE EVENTS:
Time Frame: 2 years
Description: Subjects were contacted every 3 months to inquire about adverse events, initially by phone and later by protocol mandated self-reporting via the study phone app.
Groups:
- Atorvastatin 80mg: Atorvastatin 80mg OD (optimal dose). Treatment dose will be de-escalated to 40mg based on reported adverse events.
  Atorvastatin: 80 mg OD
- Atorvastatin 40mg: Atorvastatin 40mg. Treatment dose was de-escalated to 40mg based on reported adverse events.
  Atorvastatin: 40 mg
Arm/Group | Atorvastatin 80mg | Atorvastatin 40mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/1 | 0/39
Serious Adverse Events (participants affected / at risk) | 1/40 | 1/1 | 0/39
Other Adverse Events (participants affected / at risk) | 27/40 | 1/1 | 21/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin 80mg (N=40) | Atorvastatin 40mg (N=1) | Placebo (N=39)
Elevated creatine kinase (CK) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — One subject had elevated creatine kinase on laboratory tests, without overt symptoms.
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) — One subject was hospitalized after a fall, determined to have a questionable relationship to the study drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin 80mg (N=40) | Atorvastatin 40mg (N=1) | Placebo (N=39)
Hepatitis, type unknown (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID (Infections and infestations) | 5 (5) | 0 (0) | 4 (4)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 6 (9) | 0 (0) | 3 (3)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophogeal reflux (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Cardiac disorders, other (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Elevated PSA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorder, other (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Joint range of motion decreased - foot (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral Valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - other (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Shingles (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - other (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT02603328/Prot_SAP_000.pdf